CLINICAL TRIAL: NCT02087826
Title: Study of Clinical Response to Acute Metformin By Leveraging Evaluations During a Mixed Meal Tolerance Test for Exploring Glycemia and GeneticS (SCRAMBLED EGGS)
Brief Title: Study of Clinical Response to Acute Metformin By Leveraging Evaluations During a Mixed Meal Tolerance Test for Exploring Glycemia and GeneticS
Acronym: SCRAMBLED EGGS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Instituto Carlos Slim de la Salud (Unknown); Broad Institute of MIT and Harvard (Other)
Responsible Party: Principal Investigator, Laura Natalie Brenner, Instructor in Medicine, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014P000255
Record Dates: First submitted 2014-03-12; First posted 2014-03-14 (Estimated); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Genetics; Metabolism; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Carriers of the SLC16A11 risk allele (Active Comparator): Day 1: Mixed Meal Tolerance Test
  Day 3-7: 500mg metformin, twice daily
  Day 8: Mixed Meal Tolerance Test in presence of Metformin
  Interventions: Other: Mixed Meal Tolerance Test; Drug: Metformin
- Non-carriers of the SLC16A11 risk allele (Placebo Comparator): Day 1: Mixed Meal Tolerance Test
  Day 3-7: 500mg metformin, twice daily
  Day 8: Mixed Meal Tolerance Test in presence of Metformin
  Interventions: Other: Mixed Meal Tolerance Test; Drug: Metformin

INTERVENTIONS:
Other: Mixed Meal Tolerance Test — The meal will provide a standard amount of total calories, protein, fat, and carbohydrate to each participant at both study visits. Pre-packaged and prepared food, weighed to the nearest gram, will be used.
Drug: Metformin — Metformin will be administered during this study. This medication is safely prescribed at a maximum dose of 1000 mg twice daily for the treatment or prevention of type 2 diabetes, as well as for other metabolic conditions. To minimize potential side effects of metformin (e.g., GI upset), participants will take ½ the maximum dose of this medication (500 mg twice daily) and for only 5 days. Participants will be informed of the potential side effects of metformin. They will be asked to contact study staff and discontinue the medication if symptoms are very uncomfortable.
  Other Names: Glucophage; Glumetza; Glucophage XR; Fortamet

SUMMARY:
The purpose of this research study is to examine whether specific genes (e.g. SLC16A11) affect how human beings respond to food and a medication that is commonly used to treat type 2 diabetes. The food the investigators will be studying is specially prepared to contain protein, carbohydrate, and fat. The drug the investigators are studying is metformin. The investigators hypothesize that physiological responses to the meal and to the medication will differ between carriers and non-carriers of genes associated with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or non-pregnant females
* Age 18-79
* Able and willing to give consent relevant to genetic investigation

Exclusion Criteria:

* Women who are pregnant, nursing, or at risk of becoming pregnant
* Currently taking any medications used for the treatment of diabetes
* History of liver disease and/or aspartate aminotransferase (AST) or alanine aminotransferase (ALT) more than 3 times upper limit of normal (ULN)
* Estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m2 as calculated by the Modification of Diet in Renal Disease equation
* Currently taking or intending to take during the study duration any medication known to affect glycemic parameters, such as glucocorticoids, growth hormone, or fluoroquinolones
* Contraindications to safe use of metformin, including planned radiologic or angiographic study requiring contrast within one week of the study completion
* Planned changes to any prescribed medications, specifically diuretics, during study enrollment
* Participation in any other interventional study during the study duration
* Conditions causing intestinal malabsorption, including celiac disease or a history of intestinal or gastric bypass surgery
* Dietary restrictions that would prevent consumption of a MMTT
* Objection or inability to take metformin

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1017 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Response to the Mixed Meal Tolerance Test | 2 hours after the meal
  Primary endpoint point: 2 hr glucose after the MMTT
  Secondary endpoints: 2 hr insulin after the MMTT, change in glucose, insulin, and amino acid and lipid metabolites from baseline to 60 and 120 minutes after the MMTT; change in GLP-1 concentrations from baseline to 5,10, 15, 30, 60, and 120 minutes after the MMTT; and glucose, insulin, and GLP-1 AUC over 120 minutes

SECONDARY OUTCOMES:
Response to Metformin | Day 8 of the study
  Primary endpoint: change in fasting glucose from Visit 1 to Visit 2
  Secondary endpoints: change in fasting insulin, amino acid and lipid metabolites, GLP-1, and HOMA-IR from Visit 1 to Visit 2

OTHER OUTCOMES:
Response to a Mixed Meal Tolerance Test after Metformin | 2 hours after the meal
  Primary endpoint point: 2 hr glucose after the MMTT
  Secondary endpoints: 2 hr insulin after the MMTT, change in glucose, insulin, and amino acid and lipid metabolites from baseline to 60 and 120 minutes after the MMTT; glucose, insulin, and GLP-1 AUC over 120 minutes; and intra-individual change in the above variables from Visit 1 to Visit 2

CONTACTS AND LOCATIONS:
Overall Officials: Laura N Brenner, MD, Study Director — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States